CLINICAL TRIAL: NCT07210229
Title: The Effectiveness of a Proprietary Ashwagandha Extract on Menopausal Symptoms: A Three-Arm Randomized, Double-Blinded, Placebo Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Principal Investigator, Jessie Hawkins, Primary Investigator, Nutraceuticals Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 25-08-200
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Menopausal Hot Flashes; Menopausal Women
Keywords: ashwagandha
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plant Extract 1 (Experimental): Participants in this arm will take an ashwagandha root supplement each day for 84 days.
  Interventions: Dietary Supplement: ashwagandha root
- Plant Extract 2 (Experimental): Participants in this arm will take an ashwagandha root and leaf supplement each day for 84 days.
  Interventions: Dietary Supplement: ashwagandha root and leaf
- Placebo (Placebo Comparator): Participants in this arm will take an inert placebo each day for 84 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: ashwagandha root — This substance is extracted from the root of the plant.
  Arms: Plant Extract 1
Dietary Supplement: ashwagandha root and leaf — This substance is extracted from both the root and leaves of the plant.
  Arms: Plant Extract 2
Other: Placebo — The inert placebo does not contain any of the plant matter.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of two proprietary ashwagandha extracts on symptoms of menopause and hormone levels, as compared to a placebo.

DETAILED DESCRIPTION:
Participants will take one of two extracts or a placebo every day for 84 days; outcomes of self-report menopausal symptoms collected on a trio of scales will provide information on effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness and demonstrated ability to comply with all study procedures, as well as availability for the duration of the study
* Baseline score of above-average menopause symptom levels on each of the patient reported scales: NRI-MSS (defined as 22+), the MRS scale (defined as 9+), AND 4+ on the MENQoL.
* Confirmation of presence of hot flashes
* Estridiol levels within the bottom 35% of normal ranges for their menstrual cycle phase (follicular/ovulation/luteal) as established by laboratory reference range
* Biological sex of female; gender identification of woman
* Aged 40 to 55, inclusive
* Good general health as evidenced by medical history and screening
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional month after the end of the study
* Still menstruating regularly (defined at least one period every 60 days)
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Pregnant, trying to conceive, or breastfeeding
* Hysterectomy, uterine ablation, or related procedure
* Amenorrhea
* Consumes > 8 alcoholic beverages in an average week
* Currently consumes an ashwagandha supplement or has consumed one regularly (defined as 1x week or more often) within the past 24 months
* Consumes any hormonal therapies or menopause-related supplements intended to improve symptoms in any way
* Current or recent (within 60 days) history of taking thyroid medications, hypertensive drugs, CNS depressants, diabetic medications, benzodiazepines, or immunosuppressants
* Any liver, kidney, hormonal, or cardiovascular disorder
* Known allergic reactions to any components of the intervention
* Recent dramatic weight changes (10% change in body weight in the last 6 months)
* Introducing a new investigational drug or other intervention within 60 days before the start of the study
* Any change to diet or lifestyle within 60 days before the start of the study (defined as introducing any new exercise activity, joining a gym, starting a new routine, moving to a new home, adjusting dietary habits (e.g. vegetarian, paleo, etc) or discontinuing any habits or diets.
* Any health or medical condition which, in the primary investigators opinion, may interfere with the conduct of the study

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Biological sex of woman, gender identity of female
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proprietary Menopause Symptom Scale (NRI-MSS) | days 0, 28, 56, and 84
  Nutraceuticals Research Institute's Menopause Symptom Scale is a validated self-report scale measuring symptoms across 6 domains. Scores range from 0-30, with higher scores indicating greater symptom severity.
Menopause-Specific Quality of Life (MenQoL) | days 0, 28, 56, and 84
  The MenQoL evaluates quality of life among menopausal women. Scores range from 0-8 with higher scores indicating greater symptom severity.
Menopause Rating Scale (MRS) | Days 0, 28, 56, and 84
  The MRS is a self report assessment of menopausal symptoms with scores ranging from 0-44. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Estriol | days 0, 84
  Laboratory test for estriol levels
Estradiol | days 0, 84
  Laboratory test for estradiol levels

CONTACTS AND LOCATIONS:
Locations (1):
- Nutraceuticals Research Institute, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data is available with IRB authorization and consent from all participants.